CLINICAL TRIAL: NCT00704613
Title: Planning Margin Requirements for Pediatric Radiation Oncology
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RTMRG1
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Pediatric Radiation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The planning target volume (PTV) and planning organ at risk volume (PRV) margins used for pediatric radiation therapy are empiric, and quantitative assessment of these margins is needed to improve therapy planning and delivery.

DETAILED DESCRIPTION:
Data will be gathered to develop a model to quantify the setup margin (SM) portion of the planning target volume (PTV) margin for pediatric tumor sites according to age, localization technique, treatment position, and the use of general anesthesia. Patient specific PTV and PRV margin recommendations will be developed based on the number of participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients will receive conformal or intensity-modulated radiation therapy (3D or IMRT).
* Research participant or legal guardian/representative gives written informed consent.

Exclusion Criteria:

* Unwillingness of research participant or legal guardian/representative to give written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving external beam radiation therapy at St. Jude Children's Research Hospital will be screened for participation on this research protocol based on the Inclusion Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2008-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Acquire data to develop setup margin (SM) portion of the planning target volume (PTV) margin for pediatric tumor sites according to age, localization technique, treatment position, and the use of general anesthesia. | 4 year

SECONDARY OUTCOMES:
Estimate the number of patients required to develop a patient specific PTV and RTV margin recommendations. | 4 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Merchant, DO, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org